CLINICAL TRIAL: NCT01146080
Title: Optical Coherence Tomography for EVERolimus Eluting STent (OCTEVEREST)
Brief Title: Optical Coherence Tomography for EVERolimus Eluting STent
Acronym: OCTEVEREST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Case Western Reserve University (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, GGuagliumi, MD, A.O. Ospedale Papa Giovanni XXIII
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG-001-09
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stent; everolimus eluting stent; optical coherence tomography; intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promus Element (Experimental): 21 consecutive patients with Promus Element implanted to treat coronary artery lesion
  Interventions: Device: Promus Element
- Promus (Active Comparator): 21 consecutive patients with Promus stent implanted to treat coronary artery lesions
  Interventions: Device: Promus

INTERVENTIONS:
Device: Promus Element — Promus Element implanted to treat coronary artery lesions.
  Arms: Promus Element
Device: Promus — Promus stent implanted to treat coronary artery lesions
  Arms: Promus

SUMMARY:
Compared with bare metal stents (BMS), both paclitaxel-eluting stents (PES) and sirolimus-eluting stents (SES) significantly reduce angiographic restenosis and the need for repeat revascularization in coronary arteries across a broad range of patient and lesion types. However the increased risk of very late stent thrombosis represents a major concern for patients treated with both PES and SES. Optical coherence tomography (OCT), a new imaging technique based on the back reflection of near infrared light, enables real-time, full tomographic, in-vivo visualization of coronary vessel microstructure. Struts coverage and vessel response of drug eluting stent (DES) compared to BMS are the most immediate clinical applications of OCT. Thickness of coverage and strut apposition can be quantified at micron-scale level with a resolution 10-30 times higher than conventional intravascular ultrasound (IVUS). The objective of this study OCTEVEREST (Optical Coherence Tomography for EVERolimus Eluting STent) is to evaluate the long term struts coverage and vessel wall response (abnormal intraluminal defects, strut malapposition, vessel expansions) to the PROMUS™ Everolimus Eluting Stent compared to PROMUS ELEMENT™ Everolimus Eluting Stent implanted for the treatment of stenosis in native coronaries. To investigate the completeness of struts coverage as well as the proportion of malapposed struts and the neointima characteristics, high resolution (~ 10 µ axial) intracoronary Optical Coherence Tomography (OCT) and intravascular coronary ultrasound (IVUS) will be used.

DETAILED DESCRIPTION:
This is a prospective single center clinical study designed to evaluate the long term struts coverage and vessel wall response (abnormal intraluminal defects, strut malapposition, vessel espansions) to the PROMUS™ Everolimus Eluting Stent compared to PROMUS ELEMENT ™ Everolimus Eluting Stent implanted for the treatment of stenosis in native coronaries. The difference between the two stents is in the stent platform made of a novel alloy of chromium-platinum with low strut thickness and stent crossing profile (0.042" [1.062 mm]) for PROMUS ELEMENT ™ Everolimus Eluting Stent. To investigate the completeness of struts coverage as well as the proportion of malapposed struts and the neointima characteristics, high resolution (~ 10 µ axial) intracoronary Optical Coherence Tomography (OCT) and intravascular coronary ultrasound (IVUS) will be used. The study will be carried out at Ospedali Riuniti di Bergamo, Italy with a target enrollment of consecutive 21 patients for each group receiving one or two Everolimus Eluting stents. All patients enrolled in the study will be followed to 12 months post stent placement.

PLATFORM TO BE USED PROMUS™ everolimus eluting stent. Stent sizes: 2.5 to 3.5 mm, 12 - 15 - 20 - 23 - 28 mm in lengths (according to product specifications).

PROMUS ELEMENT ™ Everolimus Eluting Stent. Stent sizes: 2.5 to 3.5 mm, 12 - 15 -20 - 23 - 28 mm in lengths (according to product specifications).

Patients presenting with a coronary artery lesion who are considered candidates for percutaneous coronary intervention and stent placement are eligible for the OCTEVEREST (Optical Coherence Tomography for EVERolimus Eluting STent)trial. Patients may have a second study lesion that can be treated with a second PROMUS™ Stent or PROMUS ELEMENT ™ Everolimus Eluting Stent.

Patients who do not meet all inclusion/exclusion criteria will not be enrolled or followed in the study. All patients who are candidates for the OCTEVEREST trial and undergo placement of the device must be consented prior to any data collection by a member of the institution's research team. All patients enrolled will be evaluated according to this protocol, regardless of sequence of treatment that ensues. More than one study lesion in different epicardial vessels may be treated in the same stage procedure. Actual study enrollment occurs following successful pre-dilatation of the study vessel, when the study device is introduced into the body. The target lesion must be able to be covered with a single stent. For diffuse lesions the total lesion length will be measured from the proximal shoulder of the most proximal lesion to the distal shoulder of the most distal lesion and should not exceed 24 mm. At 6 month follow-up, the entire stented region will be used to determine the mean lumen diameter and the percent diameter stenosis.

Optical coherence tomography (OCT) will be performed baseline and at 6 month follow up. Study site is requested to use the same OCT equipment for both procedures. The OCT procedure will be conducted according to Optical Coherence Tomography as specified by the Protocol. Optical Coherence Tomography images will be acquired at 15-30 frames per second (500 angular pixels x 250 radial pixels), from a 0.006" micro-optic core, 0.014" image wire, displayed with an inverse gray-scale lookup table, and digitally archived. The optical source used in this study has a center wavelength of 1310 nm and a bandwidth of 70 nm, providing an axial resolution of (10-12 μm in tissue with a tissue penetration of 2 mm). The transverse resolution, determined by the spot size of the sample arm beam, is 25 μm. OCT images will be analyzed by an independent Corelab (Cardialysis, Cleveland) expert in high resolution OCT analysis. An automatic analysis with novel dedicated software will be used for quantitative assessment. Interactive revision of contour appropriateness will be performed by experienced readers. In a blind fashion 10% of all sections will be re-evaluated to estimate the measurement variability (k value). The existence of malapposition will be assessed.

Angiography Angiography will be performed at baseline prior to stent placement, after stent placement, and at 6 month follow up. The Angiography procedure will be conducted according to Angiographic Core Laboratory procedure .A baseline angiography of the involved vessel will be performed in at least two near orthogonal views. Visual angiographic assessment will be used to determine if the lesion meets angiographic entry criteria. The study lesion must be free of foreshortening or vessel overlap. If angiography demonstrates that the target lesion meets study eligibility criteria, then the patient may be enrolled in the study.

Intravascular Ultrasound IVUS will be performed at the time of index procedure and at 6 month follow up. IVUS will initially be performed after successful, uncomplicated stent implantation (diameter stenosis <10%, TIMI-3 flow). Study site IS requested to use the same IVUS equipment for both procedures. IVUS will be performed on all patients according to IVUS Core. Laboratory Acquisition Protocol. Imaging will be performed with a 40 MHz Atlantis catheter (Boston Scientific), after 50- 200 mcg of intracoronary nitroglycerin. Automated motorized pullback at 0.5 mm/sec will utilized during all IVUS runs (Hi-Lab Boston Scientific). Imaging will include the edges at least 5 mm proximal and distal to the stent. The transducer will be advanced at least 10 mm distal to the distal edge of the stent(s), and a continuous, uninterrupted imaging run performed to a point at least 10mm proximal to the proximal edge of the stent(s). All IVUS studies will be archived for subsequent CoreLab analysis in DICOM format. IVUS analysis will include measurements of external elastic membrane (EEM), stent, and lumen cross-sectional areas and volumes according to the Standards for the Acquisition, Measurement, and Reporting of Intravascular Ultrasound Studies. In addition, qualitative analysis (incomplete apposition, dissections) will also be performed according to the same standards document.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has documented stable angina pectoris (Canadian Cardiovascular Society [CCS] Classification 1, 2, 3, or 4) or documented silent ischemia; or unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C)
* Patient demonstrates a left ventricular ejection fraction (LVEF) of ≥ 40% as measured prior to enrollment
* Patient understands and agrees to comply with all specified study requirements and provides written Informed Consent to this effect.

Angiographic Inclusion Criteria

* Target lesion must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥ 2.50 mm and ≤ 3,75 mm.
* Target lesion length must measure (by visual estimate) ≤ 24 mm.
* Target lesion must be in a major coronary artery or branch with visually estimated stenosis ≥ 50% and <100% with TIMI flow >1.

Exclusion Criteria:

1. General Exclusion Criteria

   * The patient has a life expectancy of less than 24 months due to another medical condition
   * Patient has a history of hypersensitivity to everolimus or paclitaxel or structurally related compounds
   * Patient exhibits cardiogenic shock (systolic pressure < 80mm Hg and PCWP > 20mm Hg or cardiac index <1.8 liters/minute/m2 or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure>80 mm Hg) for any time within 24 hours prior to index procedure
   * Patient demonstrates evidence of acute or chronic renal dysfunction (serum creatinine > 2.0 mg/dl or 177 μmol/l)
   * Planned cardiac surgery procedure ≤ 6 months post-index procedure
   * Patient demonstrates evidence of a acute myocardial infarction (eg. STEMI or enzyme elevation CK > 2X local laboratory's ULN unless CK-MB is < 2X ULN) 7)
   * Cerebrovascular accident (CVA) including stroke or TIA within previous 3 months
   * Patient demonstrates evidence of leukopenia (leukocyte count < 3.5 X 109/liter)
   * Patient demonstrates evidence of thrombocytopenia (platelet count < 100,000/mm3) or thrombocytosis (>750,000/mm3)
   * Patient is contraindicated to Aspirin (successful prior desensitization to Aspirin is not an exclusion), clopidogrel, or ticlopidine
   * Patient is currently on warfarin, or possibility of treatment with warfarin during the following 6 months post index procedure
   * Patient has been treated with paclitaxel, everolimus or other chemotherapeutic agents within 12-months prior to planned index procedure
   * Anticipated treatment with paclitaxel, everolimus or oral rapamycin during any period in the 6-months after the index procedure
   * Known allergy to stainless steel
   * Female or male with known intention to procreate within 3 months after the index procedure (due to the exposure to paclitaxel and unknown affect it may have on the fetus)
   * Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the 9 months post index procedure
   * Patient that in the opinion of the investigator is not clinically appropriate for OCT evaluation.
2. Angiographic Exclusion Criteria

   * Evidence of thrombus of the study vessel, based on angiography or IVUS
   * Study lesion is totally occluded (TIMI flow ≤ 1) either at baseline or before predilatation
   * Study lesion, or the study vessel proximal to the study lesion is moderately or severely calcified, by visual estimate
   * Study lesion is ostial in location (within 5.0 mm of vessel origin)
   * Study lesion involving arterial segments with highly tortuous anatomy or where lesion is located within or distal to a >60 degree bend in the vessel
   * Study lesion involves a bifurcation with a diseased (>50% stenotic) branch - Left main coronary artery disease (stenosis >50%) whether protected or unprotected
   * Target lesion length > 24 mm, based on visual estimate by operator
   * Target vessel diameter > 3.75 mm, based on visual estimate by operator
   * Target vessel diameter < 2.5 mm based on visual estimate by operator
   * Pre-treatment of the target lesion (excluding predilation) with another interventional device.
   * Target lesion is restenotic from previous intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of stent struts uncovered at 6 months as measured by OCT | 6 months
  The proportion of stent struts uncovered by endothelial tissue will be determined by measuring the number of exposed struts, defined as a measured neointimal hyperplasia (NIH) thickness less than 10 μm, at 0.5 mm cross section analysis, divided by the total number of stent struts. This analysis shall be performed using a dedicated software, as assessed by OCT core lab at 6 month follow up.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1,6,12,24 months
  including any cardiac death, myocardial infarction (Q wave and non Q wave MI) and target vessel revascularization at 6 month follow-up. All specific components of MACE will be summarized. MACE shall be assessed at discharge (or within 7 days post index procedure, whichever comes first), 1, 6, 12 and 24 month follow up
Stent Thrombosis rate through 24 months | 24 months
  based on the Academic Research Consortium - ARC definitions (definite, probable or possible). Stent thrombosis shall be considered subacute stent thrombosis if it occurs < 30 days after stenting; late stent thrombosis if it occurs > 30 days and ≤ 1 year after index stenting and very late stent thrombosis if it occurs > 1 year and ≤ 2 years after index procedure.
Target Lesion Revascularization | 24 months
  Any repeat revascularization procedure (percutaneous or surgical) of the original target lesion site, which includes the stented plus edge (typically 5 mm proximal and distal to the stent) segments
QCA parameters: | 6 months
  mean lumen diameter, acute gain, late loss through 6 months, and binary restenosis (≥ 50% diameter stenosis) rate at 6 months follow-up as determined by Quantitative Coronary Angiography
Additional OCT parameters | 6 months
  Neointimal thickness at every 0.5 mm sections- mean and max, proportion of Low Intensity Parastrut Material, number and size of abnormal intraluminal masses related to malapposed struts, neointima characterization at 6 months follow-up
IVUS parameters | 6 months
  including neointimal area volume, stent and area volumes, stent apposition, and percent net volume obstruction at 6 months as determined by intravascular ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Cardiovascular Department Ospedali Riuniti di Bergamo, Bergamo, BG, Italy

REFERENCES:
- [Derived] Guagliumi G, Capodanno D, Ikejima H, Bezerra HG, Sirbu V, Musumeci G, Fiocca L, Lortkipanidze N, Vassileva A, Tahara S, Valsecchi O, Costa MA. Impact of different stent alloys on human vascular response to everolimus-eluting stent: an optical coherence tomography study: the OCTEVEREST. Catheter Cardiovasc Interv. 2013 Feb;81(3):510-8. doi: 10.1002/ccd.24374. Epub 2012 May 2. PMID 22431208